CLINICAL TRIAL: NCT01415479
Title: Trial of a Computer-Based Presentation of Quantitative Information About Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Peter Schwartz, Assistant Professor of Medicine, Indiana University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: CCCDA-10-085-01-A; VFR-320-A (Other Grant/Funding Number: IU Health Values Fund)
Record Dates: First submitted 2011-08-02; First posted 2011-08-12 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Colonic Neoplasms
Keywords: Colon cancer; Screening; Decision-making
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Quantitative (Experimental): Subjects view:
  1. Computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy, sigmoidoscopy, or stool testing. Includes a video from the American Cancer Society.
  2. Computer-based presentation providing quantitative information regarding (a) the lifetime average probability of getting CRC or dying from it, (b) the reduction in mortality provided by undergoing regular screening with colonoscopy, and (c) the reduction in mortality provided by undergoing regular screening with fecal immunochemical testing (FIT)
  Interventions: Behavioral: Control; Behavioral: Quantitative
- Default (Experimental): Subjects view:
  1. Computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy, sigmoidoscopy, or stool testing. Includes a video from the American Cancer Society.
  2. Computer-based presentation that encourages subjects who are unwilling to undergo colonoscopy or are unsure about whether to undergo screening to get tested with Fecal Immunochemical Testing (FIT).
  Interventions: Behavioral: Control; Behavioral: Default
- Quantitative + Default (Experimental): Subjects view:
  1. Computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy, sigmoidoscopy, or stool testing. Includes a video from the American Cancer Society.
  2. Computer-based presentation providing quantitative information regarding (a) the lifetime average probability of getting CRC or dying from it, (b) the reduction in mortality provided by undergoing regular screening with colonoscopy, and (c) the reduction in mortality provided by undergoing regular screening with fecal immunochemical testing (FIT)
  3. Computer-based presentation that encourages subjects who are unwilling to undergo colonoscopy or are unsure about whether to undergo screening to get tested with Fecal Immunochemical Testing (FIT).
  Interventions: Behavioral: Control; Behavioral: Quantitative; Behavioral: Default
- Control (Active Comparator): Subjects view a computer-based presentation regarding colorectal cancer (CRC) and available screening tests for CRC, primarily a video produced by the American Cancer Society.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — Computer-based presentation regarding colorectal cancer (CRC) and screening for CRC with colonoscopy, sigmoidoscopy, or stool testing. Includes a video from the American Cancer Society.
Behavioral: Quantitative — Computer-based presentation providing quantitative information regarding (a) the lifetime average probability of getting CRC or dying from it, (b) the reduction in mortality provided by undergoing regular screening with colonoscopy, and (c) the reduction in mortality provided by undergoing regular screening with fecal immunochemical testing (FIT)
  Arms: Quantitative; Quantitative + Default
Behavioral: Default — Computer-based presentation that encourages subjects who are unwilling to undergo colonoscopy or are unsure about whether to undergo screening to get tested with Fecal Immunochemical Testing (FIT). This is labeled the "Default" intervention since it attempts to shift the "default" choice from "no screening" to FIT.
  Arms: Default; Quantitative + Default

SUMMARY:
Fifty thousand people die from colorectal cancer (CRC) every year, making it the second leading cause of death from cancer in the United States. And although there are multiple screening tests that reduce the morbidity and mortality of this disease, less than 60% of eligible individuals are up to date with recommended screening.

One of the challenges to improving screening is helping patients understand the range of approved tests, including colonoscopy, sigmoidoscopy, and stool testing (such as fecal immunochemical testing (FIT)). Patients rarely consider all their options, partly due to the limited time they have to learn about them during busy doctor's visits.

Computer-based presentations, including decision aids, are a promising tool for improving patient understanding in this and other areas, by giving patients significant amounts of information.

But there are important questions about how to design such presentations, including whether they should provide quantitative data about the risks and benefits of screening. Some experts feel that these numbers and graphs are necessary for fully informed decision-making, while others are concerned that they may confuse patients or dissuade them from screening.

The investigators have created and pilot tested a computer-based presentation of quantitative information about CRC screening. The investigators found that subjects who viewed the program in a non-healthcare setting exhibited significantly increased interest in screening. In addition, the investigators tested a version of the program that includes a "nudge" towards stool testing with FIT, as a way of encouraging individuals who are confused to undergo some form of screening. In our testing, receiving the nudge was associated with a significant increase in interest in FIT.

The investigators now seek to conduct a randomized, controlled study of our computer-based presentation with Clarian patients who are due for CRC screening. All subjects will first view a general video about CRC screening and then will be randomly placed into four groups (using a 2x2 design), to receive quantitative information (or not), and a nudge towards FIT (or not).

The results will determine whether a presentation of quantitative information can increase patient understanding, quality of decision-making, and uptake of CRC screening. The results will serve as pilot data for a larger, externally funded study of the effect of individualized ("personalized") quantitative information in this area

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years old
* No colonoscopy performed in last 10 years, sigmoidoscopy in last 5 years or fecal occult blood testing (including FIT) in last 1 year, and
* Upcoming appointment with primary care physician at three primary care sites of IU Health (previously sites of the Methodist Medical Group (MMG)): Internal Medicine and Pediatrics Fishers, Family & Internal Medicine South, or Family & Internal Medicine East Washington.

Exclusion Criteria:

* Undergoing workup for symptoms consistent with colon cancer, such as weight loss or rectal bleeding
* Diagnosis or medical history conferring elevated risk for CRC including previous polypectomy or colon cancer, inflammatory bowel disease, certain inherited syndromes, or a significant family history of CRC, or
* Inability to speak English and to fill out a questionnaire written in English.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Intention to undergo CRC screening in the next six months | Day 1: Immediately before and after viewing intervention (at the same visit)
  Multiple choice question assessing subject's interest in getting a colon screening test in the next 6 months (choices: definitely, probably, may or may not, probably not, or definitely not).

SECONDARY OUTCOMES:
Preferred CRC screening test | Day 1: Immediately before and after viewing intervention (at the same visit)
  Multiple choice question: which colon test the subject would choose if he or she was having one (choices: stool test, colonoscopy, other, or don't know).
Knowledge of CRC risk and the benefit of CRC screening | Day 1: Immediately before and after viewing intervention (at the same visit)
  8 True/False questions and 4 Multiple choice questions
Decision conflict | Day 1: Immediately before and after viewing intervention (at the same visit)
  Decision Conflict Scale
Completion of CRC screening | 6 months post-intervention
  Completion of colonoscopy, fecal immunochemical testing (FIT), or other CRC screening test, based on personal report and medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Schwartz, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Health, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Rager JB, Althouse S, Perkins SM, Schmidt KK, Schwartz PH. Measuring the Impact of Quantitative Information on Patient Understanding: Approaches for Assessing the Adequacy of Patient Knowledge about Colorectal Cancer Screening. MDM Policy Pract. 2022 Nov 25;7(2):23814683221140122. doi: 10.1177/23814683221140122. eCollection 2022 Jul-Dec. PMID 36452315
- [Derived] Schwartz PH, Perkins SM, Schmidt KK, Muriello PF, Althouse S, Rawl SM. Providing Quantitative Information and a Nudge to Undergo Stool Testing in a Colorectal Cancer Screening Decision Aid: A Randomized Clinical Trial. Med Decis Making. 2017 Aug;37(6):688-702. doi: 10.1177/0272989X17698678. Epub 2017 Apr 11. PMID 28398836